CLINICAL TRIAL: NCT05475145
Title: Resin-based Sealing vs Resin-modified Glass Ionomer Cement for Treatment of Occlusal Dentin Caries in Primary Molars
Brief Title: Sealing of Occlusal Dentin Caries in Primary Molars.
Acronym: SealCar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mats Bågesund (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Mats Bågesund, Associate Professor, Assistant Professor, Senior Consultant Specialist in Pediatric Dentistry, Region Östergötland
Organization: Region Östergötland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/297-31; #7-15-19, #7-16-7 (Other: Public Dental Service Östergötland); SPF2018 (Other: Swedish Society of Pediatric Dentistry); #565531, #666761, #862781 (Other: FORSS - Medical Research Council of South-East Sweden.)
Record Dates: First submitted 2022-06-17; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Caries; Dentin; Fissure, Dental; Dental Caries in Children; Glass Ionomer Cement; Fissure Sealants
Keywords: fissure sealant; dental atraumatic restorative treatment; deciduous teeth; glass ionomer cement; Dental Caries in Children
MeSH Terms: conditions — Dental Fissures

STUDY DESIGN:
Intervention Model Description: Non-blinded randomized split-mouth longitudinal 3 year follow up study.
Masking Description: We consider it not possible to mask för participant or care provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child (Experimental): Each patient receives treatment of dental caries in two primary molars using two diffferent methods - Resin based sealing [RBS] or Glassionomer cement [GIC].
  Interventions: Procedure: Resin based sealing [RBS]

INTERVENTIONS:
Procedure: Resin based sealing [RBS]
  Other Names: Glassionomer cement [GIC].

SUMMARY:
BACKGROUND A simple method for arresting dentin caries with a tight seal of the cavity would exclude the need for injection and excavation, reduce the risk for dental fear and possibly postpone or eliminate the need for further treatment.

AIM The aim is to evaluate success-rate and children's subjective experience of resin-based sealing (RBS) and resin-modified glass ionomer cement (GIC) for treatment of occlusal dentin caries in primary molars.

DESIGN Children aged 2-9 years will be recruited to undergo RBS- or GIC-treatment treatment for occlusal dentin caries in primary molars. A parent will answer the Short Form of Children's Fear Survey (CFSS-DS; parental version). No excavation but etching with 38% phosphoric acid will precede RBS. Topical and local anaesthesia and excavation with high speed bur will precede GIC. Time for treatment will be estimated. The children will rank their experience of each treatment on a 7-grade face scale. The dentist will evaluate the child's experience, cooperation and the overall experience of the treatment on a four-grade scale. The treatment will be evaluated as "without remark" or "defective" after 3, 6, 12, 24 and 36 months. For statistical analysis the Chi-2-test, Wilcoxon-Signed-Rank-test and Paired t-test will be used.

DETAILED DESCRIPTION:
BACKGROUND A simple method for arresting dentin caries with a tight seal of the cavity would exclude the need for injection and excavation, reduce the risk for dental fear and possibly postpone or eliminate the need for further treatment.

AIM The aim is to evaluate success-rate and children's subjective experience of resin-based sealing (RBS) and resin-modified glass ionomer cement (GIC) for treatment of occlusal dentin caries in primary molars.

DESIGN Up to 300 children aged 2-9 years will be recruited to undergo RBS- or GIC-treatment treatment for occlusal dentin caries in primary molars. A parent will answer the Short Form of Children's Fear Survey (CFSS-DS; parental version). No excavation but etching with 38% phosphoric acid will precede RBS. Topical and local anaesthesia and excavation with high speed bur will precede GIC. Time for treatment will be estimated. The children will rank their experience of each treatment on a 7-grade face scale. The dentist will evaluate the child's experience, cooperation and the overall experience of the treatment on a four-grade scale. The treatment will be evaluated as "without remark" or "defective" after 3, 6, 12, 24 and 36 months. For statistical analysis the Chi-2-test, Wilcoxon-Signed-Rank-test and Paired t-test will be used.

ELIGIBILITY:
Inclusion Criteria:

• primary occlusal dentin caries in two primary molars

Exclusion Criteria:

* Language problems or disabilities
* Less than 3 years until expected exfoliation
* Hypomineralization
* Previous filling or dentin caries
* Carious cavity >1/3 of occlusal surface
* Unable to cooperate
* Appearing caries or filling (on studied tooth) not originating from the studied cavity
* Tooth exfoliating before end of study
* Leaving Public dental service or moving out of the region during follow up period

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Treatment success without defects after 3 years | 3 years. Evaluation will be performed at each follow up visit - that is after 3 months, 6 months, 12 months ´, 24 months and after 36 months. Registration of possiblöe defects will be performed atv ech visit for each patient for each of the used methods.
  Percentage of treatments (for each of the studied groups) without defects during the 3-year follow up period

SECONDARY OUTCOMES:
Patient preferance | 3 years. From inclusion of first patient until the two treatments have been performed in each of the included children.
  Comparing patiens´experience on a 7-grade face-scale (Bieri et al.1990) of the two treatments
Dentist´s preferance | 3 years. From inclusion of first patient until the two treatments have been performed in each of the included children.
  Comparing the dentists preferance of the two tretaments methods on a four grade rank-scale from "very bad" to "very good".
Time used for the treatment | 3 years. From inclusion of first patient until the two treatments have been performed in each of the included children.
  Evaluating time used for each of the two different treatment methods - measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mats A Bågesund, PhD,AssProf, Study Director — Linkoeping University

IPD SHARING:
Plan to Share IPD: No
Results will be published on group level and data possible to connect to an individual person will not be presented.

REFERENCES:
- [Derived] Bagesund M, Olson AC, Chizarie S, Omanovic M, Zuber A, Hultquist AI. Resin-based sealing vs resin-modified glass-ionomer filling for treatment of occlusal cavitated dentine caries lesions in primary molars - a multi-center randomized controlled split-mouth 3-year follow-up clinical trial. Eur Arch Paediatr Dent. 2026 Jan 10. doi: 10.1007/s40368-026-01161-7. Online ahead of print. PMID 41520098